CLINICAL TRIAL: NCT02506673
Title: The Effect of Audiovisual Aids on Perioperative Stress Response, Pain and Overall Experience - a Randomized Controlled Pilot Study
Brief Title: Audiovisual Aid Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-394
Record Dates: First submitted 2015-07-02; First posted 2015-07-23 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: Stress, Psychological
Keywords: Audiovisual Aids; Perioperative Period; Anxiety
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedation only with skin conductance monitor (Active Comparator): Patients will receive traditional sedation with 2 mg of midazolam on arrival in the OR. Patients in this group will wear the skin conductance monitor to measure changes in levels of sympathetic discharge.
  Interventions: Drug: Midazolam; Device: Skin Conductance Monitor
- Sedation & audiovisual aids with skin conductance monitor (Experimental): Prior to surgery, patients will be asked to wear audiovisual equipment (Zeiss, Cinema ProMED) in the holding area. Patients in this group will also receive 2 mg of midazolam on arrival in OR. Patients in this group will also wear the skin conductance monitor to measure changes in levels of sympathetic discharge.
  Interventions: Device: Zeiss, Cinema ProMED (audiovisual equipment); Drug: Midazolam; Device: Skin Conductance Monitor

INTERVENTIONS:
Device: Zeiss, Cinema ProMED (audiovisual equipment)
  Arms: Sedation & audiovisual aids with skin conductance monitor
Drug: Midazolam
Device: Skin Conductance Monitor

SUMMARY:
Little is known about perioperative stress responses and possible anxiety mitigating factors like audiovisual aids or IV sedation. Most studies use surrogate markers and retrospective questionnaires, and are not based on real-time gathered data. Skin conductance measurements allow the sympathetic discharge to be evaluated down to fractions of a second and enable us to continuously monitor stress responses as skin conductance responses/per second during the perioperative management. In our study, the investigators propose to examine the effect of personal audiovisual equipment (audio/video goggles) on perioperative stress, pain, and overall experience in patients undergoing ambulatory meniscectomy under spinal anesthesia. Patients will be randomly assigned to either receive traditional sedation or light sedation in addition to audiovisual equipment. The investigators hope to determine outcome estimates of the use of this equipment on stress levels using skin conductance measurements, request for further sedation, postoperative pain levels and analgesic consumption, time to discharge readiness, and overall patient satisfaction, and collect thus far unavailable data on the stress response to perioperative stresses (such as IV insertion and spinal placement) in order to allow for power analyses for future studies.

DETAILED DESCRIPTION:
PLEASE NOTE: After conducting the interim analysis and plotting the skin conductance data, we have determined that the graphs are not consistent enough to draw any conclusions. Given the technical difficulties we have encountered with the Med-Storm Stress Detector, as well as the labor intensity associated with it, we have decided that we will no longer use it from patient 14 on. We will not mark the time points and hand movements described in the protocol, as this data was used to understand the skin conductance data. We will continue to enroll patients to complete this pilot/exploratory study, as the other secondary outcomes--in particular, the surveys--could provide valuable information.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary, ambulatory, arthroscopic meniscectomy under spinal anesthesia

Exclusion Criteria:

* Patients with psychiatric disease and those on antidepressants
* Contraindications to spinal anesthesia or allergy to study medication
* Age < 18 years
* Patients with audiovisual impairments
* Patients with inability to communicate in English or understand the study requirements
* Chronic pain patients +/- opioid use
* Patients with (neuro)dermatoses encompassing the hand
* Patients with pacemakers
* Patients with diabetes or known neuropathic disease
* Patients with a history of epilepsy or seizure disorder
* Patients with a history of claustrophobia
* Patients with a history of epilepsy
* Patients with prior history of epilepsy or seizure disorder
* Patients undergoing a revision or open procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros G. Memtsoudis, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery (HSS), New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedation Only With Skin Conductance Monitor: Patients will receive traditional sedation with 2 mg of midazolam on arrival in the OR. Patients in this group will wear the skin conductance monitor to measure changes in levels of sympathetic discharge.
  Midazolam
  Skin Conductance Monitor
- Sedation & Audiovisual Aids With Skin Conductance Monitor: Prior to surgery, patients will be asked to wear audiovisual equipment (Zeiss, Cinema ProMED) in the holding area. Patients in this group will also receive 2 mg of midazolam on arrival in OR. Patients in this group will also wear the skin conductance monitor to measure changes in levels of sympathetic discharge.
  Zeiss, Cinema ProMED (audiovisual equipment)
  Midazolam
  Skin Conductance Monitor
Period: Overall Study
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Skin Conductance Response
Description: Primary outcome will be number of skin conductance responses per second (SCR/sec) and amplitude of skin conductance responses averaged over time in 5 minute intervals and at key time points such before, during and after insertion of an IV, discussion with surgeon, anesthesiologist, immediately before leaving the holding area, immediately after entering the OR, during application of monitors, before and after administration of sedatives, before, during and after spinal insertion, incision, immediately prior to leaving the OR, after arrival at PACU and monitors are placed, before discharge from the PACU.
Time Frame: Measured in 5 minute intervals, from holding area until PACU discharge.
Population: We had planned to use the Med-Storm Stress detector to measure skin conductance throughout the procedure until discharge. However, due to repeated technical difficulties with the device and inconclusive data from an analysis of a small number of patients data collection was stopped. No data are presented here.
Measure: Mean (Standard Deviation); unit: skin conductance responses per second
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
skin conductance responses per second | NA (NA) — Due to repeated technical difficulties with the device and inconclusive data from the analysis, the data collection was stopped. There is no data to be presented here. | NA (NA) — Due to repeated technical difficulties with the device and inconclusive data from the analysis, the data collection was stopped. There is no data to be presented here.

2. Secondary Outcome: Beats Per Minute (BPM)
Description: The change in heart rate from holding area until PACU discharge.
Time Frame: Measured from preop to postop
Population: Baseline has the heart rate number but analysis for intraop and postop is the change of the variable. Some patients were discharge earlier
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
Beats Per Minute
  BPM Baseline | 71.7 (10.2) | 66.8 (8.7)
  BPM change Intraop | 17 (27) | 17 (11)
  BPM change Postop: number analyzed (Participants) | 13 | 12
  BPM change Postop | 2 (10) | -6 (14)

3. Secondary Outcome: Systolic and Diastolic Blood Pressure
Description: The maximum change in postoperative systolic and diastolic blood pressure from holding area until PACU discharge.
Time Frame: Measured from preop to postop
Population: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for baseline, intra op and post op was recorded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 013 | 013
mmHg
  DBP Baseline | 82.8 (12.7) | 79.6 (9.5)
  DBP change intraop | 3 (8) | 2 (7)
  DBP change postop: number analyzed (Participants) | 013 | 012
  DBP change postop | -2 (11) | -4 (6)
  SBP Baseline | 135.3 (14.5) | 129.2 (15.1)
  SBP change intraop | 7 (10) | 7 (14)
  SBP change postop: number analyzed (Participants) | 013 | 012
  SBP change postop | -8 (13) | -2 (15)

4. Secondary Outcome: Respiratory Rate
Description: The maxmimum change in postoperative respiratory rate from holding area until PACU discharge.
Time Frame: Measured from preop to postop
Population: Some data was not available for all participants due to equipment not working or due to early discharge
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 013 | 013
breaths/minute
  RR Baseline | 17.2 (2.2) | 16.9 (1.7)
  RR change intraop: number analyzed (Participants) | 12 | 13
  RR change intraop | 5 (12) | 4 (4)
  RR change postop: number analyzed (Participants) | 5 | 7
  RR change postop | -1 (3) | 1 (5)

5. Secondary Outcome: Number of Patients Who Requested Additional Sedation
Description: Number of patients who requested additional sedative medication in the operating room.
Time Frame: In the operating room
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
Participants | 5 | 3

6. Secondary Outcome: Pain Numerical Rating Scale (NRS) Levels
Description: Pain scores at rest will be collected from patients using the numerical rating scale (NRS), which asks patients to report their level of pain on a scale from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain. NRS levels in holding area, PACU until discharge from the PACU and one day after surgery, postop day 1.
Time Frame: Holding area, Postop (PACU, 30 minutes after arrival to PACU and POD1)
Population: Holding area, PACU arrival, 30 minutes after arrival to PACU and POD1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 013 | 013
units on a scale
  Holding area | 1.9 (1.6) | 2.2 (1.4)
  PACU arrival: number analyzed (Participants) | 013 | 012
  PACU arrival | 0 (0) | 0 (0)
  30 minutes after arrival to PACU: number analyzed (Participants) | 013 | 012
  30 minutes after arrival to PACU | 0.6 (2.2) | 0 (0)
  POD1: number analyzed (Participants) | 013 | 010
  POD1 | 2.5 (1.7) | 2.1 (1.5)

7. Secondary Outcome: Narcotic Consumption
Description: Narcotic consumption "intraop", "postop" and "POD1"
Time Frame: Preop until 24 hours after surgery (holding area until POD 1)
Population: POD1 - 13 patients from the AVA group were analyzed due to early discharge.
Measure: Mean (Standard Deviation); unit: oral morphine equivalents mg
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
oral morphine equivalents mg
  OME mg Intraop | 2.3 (8.3) | 3.5 (12.5)
  OME mg Inpatient postop | 9.8 (6) | 10.8 (5)
  OME mg POD1 | 11.0 (9.9) | 11.5 (12.3)

8. Secondary Outcome: State-Trait Anxiety Inventory Questionnaire (STAI)
Description: Questionnaire to measure state anixety levels based on a 4-point likert scale and consists of 40 questions. The questionnaire measures two types of anxiety: state anxiety and trait anxiety. State anxiety relates to anxiety about an event, while trait anxiety in anxiety level as a personal characteristic. Scores can range from 20 to 80 and higher scores correlate with more anxiety.
Time Frame: holding area and PACU
Population: 4-point likert scale and consists of 40 questions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
score on a scale
  STAI-State in holding area | 33.5 (11.4) | 32.3 (7)
  STAI-Trait in holding area | 33.4 (8.9) | 31.8 (6.0)
  STAI-State in PACU: number analyzed (Participants) | 11 | 12
  STAI-State in PACU | 26.1 (2.6) | 27.1 (5.2)
  STAI-Trait in PACU: number analyzed (Participants) | 12 | 11
  STAI-Trait in PACU | 32.3 (9.2) | 32.8 (9.4)

9. Secondary Outcome: Heidelberg Peri-anaesthetic Questionnaire
Description: The questionnaire consists of 38 questions assessing perioperative satisfaction about five identified themes: trust and atmosphere; fear; discomfort; treatment by personnel; and information and waiting. The questions are rated on a 4-point Likert scale ranging from 0 (unimportant to me) to 3 (very important to me). Higher scores indicate higher levels of satisfaction. Patient satisfaction (Heidelberg Peri-Anaesthetic Questionnaire) in PACU upon spinal resolution.
Time Frame: At PACU upon spinal resolution.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 12
score on a scale | 97.2 (14.0) | 98.9 (9.5)

10. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: The client satisfaction questionnaire (CSQ-8) is a standardized satisfaction measure and was used to collect patient feedback on the audio visual devices. Response options differ, but all are on a 4-point scale. Scores range from 8 to 32, with higher values indicating higher satisfaction. Patient feedback (CSQ8) in PACU upon spinal resolution provider feedback (form sent to providers at end of surgery day)
Time Frame: PACU upon spinal resolution
Population: This questionnaire was only administered to patients who used the audio-visual aids
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 0 | 12
scores on a scale |  | 31.5 [27 to 32]

11. Secondary Outcome: Number of Providers That Were Satisfied With Their Experience With the Audio-visual Aids
Description: Anesthesia providers were asked to provide feedback on their experience with the audio-visual aids when the randomization was for the use of the device. This was collected upon surgery end.
Time Frame: Sent to providers at end of surgery.
Population: Providers were only asked to provide feedback on the equipment when used by patients in the audiovisual aid group upon surgery end.
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 0 | 011
Participants |  | 07

12. Secondary Outcome: Request of Sedation/Termination of AVA
Description: Request of Sedation/Termination of AVA (After consent has been obtained until spinal resolution in the recovery room, average of 6 hours)
Time Frame: From consent until spinal resolution (avg 6 hs)
Population: This outcome is only providing findings for subjects that has sedation and audiovisual aids with skin conductance monitor. It does not pertain to subjects that had sedation without the AVA.
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 0 | 13
Participants
  Number of Participants (AVA Randomization) |  | 13
  Request of Sedation/Termination of AVA |  | 13

13. Secondary Outcome: Number of Participants With Complications
Description: The percentage of patients who experienced complications (headache, transient neurologic symptoms, nausea and vomiting, ...)
Time Frame: Intraoperatively and in the recovery room, average of 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
Number analyzed (Participants) | 13 | 13
Participants
  Incidence of Complication Intraop | 0 | 0
  Incidence of Complication PACU | 0 | 0

ADVERSE EVENTS:
Time Frame: Data will be collected on the day of surgery in the holding area, during the procedure, in the PACU until discharge, and on post-operative day 1, 6 months and 1 year; however no patients experiences any adverse events
Arm/Group | Sedation Only With Skin Conductance Monitor | Sedation & Audiovisual Aids With Skin Conductance Monitor
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT02506673/Prot_SAP_000.pdf